CLINICAL TRIAL: NCT04006873
Title: A Randomised Crossover Pilot Study of the Effects of Tezacaftor/Ivacaftor and Ivacaftor on Gastrointestinal Function Using Magnetic Resonance Imaging Parameters in People With Cystic Fibrosis
Brief Title: Gut Imaging for Function & Transit in Cystic Fibrosis Study 2
Acronym: GIFT-CF2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Nottingham University Hospitals NHS Trust (Other)
Collaborators: Vertex Pharmaceuticals Incorporated (Industry); Cystic Fibrosis Foundation (Other); Cystic Fibrosis Trust (Other); University of Nottingham (Other); Nottingham University Hospitals Charity (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: 18RM039
Record Dates: First submitted 2019-07-02; First posted 2019-07-05 (Actual); Last update posted 2023-05-24 (Actual); Status verified 2023-05

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — tezacaftor, ivacaftor drug combination; tezacaftor; ivacaftor; Exercise

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Tezacaftor/Ivacaftor in combination with Ivacaftor (Active Comparator): A film-coated tablet containing 100mg tezacaftor and 150mg ivacaftor will be taken in the morning.
  A film-coated tablet containing 150mg ivacaftor will be taken in the evening.
  Participants will take these tablets for 28 days.
  All tablets are licensed for use in the EU.
  Interventions: Drug: Tezacaftor/Ivacaftor + Ivacaftor
- Placebo (Placebo Comparator): A visually matched placebo to the active drugs will be taken in the morning and in the evening for 28 days.
  Interventions: Drug: Placebo oral tablet

INTERVENTIONS:
Drug: Tezacaftor/Ivacaftor + Ivacaftor — As per description in arms.
  Other Names: VX-661 100mg / VX-770 150mg active tablets; VX-770 150mg active tablets
  Arms: Tezacaftor/Ivacaftor in combination with Ivacaftor
Drug: Placebo oral tablet — As per description in arms
  Other Names: Matching placebo tablets
  Arms: Placebo

SUMMARY:
People with Cystic Fibrosis (CF) have problems digesting their food properly. More than 8 in 10 people with CF must take medication to assist their digestion. In spite of this, complications such as bowel blockage occur.

Finding out how already licenced drugs for CF work in the gut is the first step in repurposing medications. Tezacaftor/Ivacaftor with Ivacaftor is a drug combination which corrects the basic defect in CF an has shown improvements on lung function.

The purpose of this study is to evaluate, using Magnetic Resonance Imaging (MRI) and patient-reported outcomes, whether Tezacaftor/Ivacaftor with Ivacaftor has an effect on improving gastrointestinal problems in CF.

DETAILED DESCRIPTION:
This is a small pilot study to compare the effects of active drug (Tezacaftor/Ivacaftor with Ivacaftor) on the gut in people with CF.

Participants will be randomised to take active drug or matched placebo for 28 days then switch to the alternate drug after a 28 day washout period. Before participants commence treatment, they will have blood pressure and baseline blood tests.

Participants will attend once per treatment period for MRI scanning at the Sir Peter Mansfield Imaging Centre, after an overnight fast. On this day, participants will be asked to withhold any medicines directly altering bowel habit such as laxatives. They will continue to take pancreatic enzyme replacement therapy and other medications for CF.

The Investigators will use the same MRI protocol as described in GIFT-CF (NCT03566550). Participants will have their first MRI scan fasted. After the first scan, they will eat a first standardised meal . They will then have 7 MRI scans at half hourly intervals and 3 MRI scans at hourly intervals. Participants will be given a second standardised meal after their ninth MRI scan. Each MRI scan will last approximately 15 minutes. After each MRI scan, participants will complete a validated gastrointestinal symptom questionnaire (Gastrointestinal Symptom Rating Scale). In between scans, participants will have access to an adjacent room with Wifi and television access.

During the day, participants will have their lung function, blood pressure and blood tests taken. They will also provide a sputum and stool sample.

Infection control requirements mean that only 1 participant will attend for MRI scanning per day.

***Amendment to study due to COVID-19*** From mid-March 2020, all face to face clinical research in the UK has been suspended (apart from studies directly related to the COVID-19 pandemic). Patients in the GIFT-CF 2 trial who had not yet completed the full trial protocol were therefore unable to continue. Funding for SymkeviTM (tezacaftor/ivacaftor and ivacaftor) in the UK was announced at the end of 2019 and some of the trial participants, who have not completed GIFT-CF 2, may be prescribed SymkeviTM by their CF team. It will therefore not be possible for them to complete the placebo controlled cross-over trial, once COVID restrictions are eased. We plan to mitigate the effects of COVID-related disruption by ensuring all trial participants have had the full, protocol-defined, scan sequence both on and off SymkeviTM. When restrictions are eased, we will invite participants who have been prescribed SymkeviTM by their CF centre to attend for scanning, if they have not previously had an "on treatment" scan. We will follow the same scanning protocol. We will ensure that adherence to SymkeviTM is good and they have received at least 21 days of treatment (as specified in the trial protocol). Our primary analysis will be on the patients who completed the trial per protocol but we will present a secondary analysis on all 12 patients, comparing outcome measures on SymkeviTM with their outcome measures previously recorded at baseline (off treatment). The personnel interpreting the MRI scans will be blind to whether they were performed on or off SymkeviTM - reducing the probability of observer bias.

***Post hoc analysis*** For participants who are invited for an open-label "on treatment" MRI scan day, the statistical analysis will involve a comparison between their pre-treatment MRI scans and the open-label scan. The researcher analysing the images will remain blinded. Statistical analysis for these participants will be a comparison between their pre-treatment scan and open-label on-treatment scan. Motility outcomes will not be analysed as the specific MR sequencing was adapted to focus on the terminal ileum in the cross-over trial, whilst in the pre-treatment scans, the motility was across the whole small bowel.

ELIGIBILITY:
Inclusion Criteria:

* capacity to consent, or to understand the requirements of the study where parental consent is needed
* confirmed diagnosis of CF, either by sweat test or genetic testing. Tezacaftor/Ivacaftor is indicated only for patients homozygous for the commonest CF mutation - p.Phe508del and so we will enrol only CF patients with this genotype

Exclusion Criteria:

* currently taking CFTR modulator drug
* Contra-indication to use of Tezacaftor/Ivacaftor
* Measurement of FEV1 <40% predicted using Global Lung Initiative criteria, according to clinical records, as participants will be required to perform a series of 10 second breathholds throughout MRI scanning
* Contra-indication to MRI scanning, such as embedded metal, pacemaker.
* Pregnancy
* Unable to stop medications directly prescribed to alter bowel habit, such as laxatives or anti-diarrhoeals, on the study day
* Previous resection of any part of the gastrointestinal tract apart from appendicectomy or cholecystectomy. Surgical relief of meconium ileus or DIOS will be permitted unless clinical records show excision of intestine >20cm in length.
* Intestinal stoma
* Diagnosis of inflammatory bowel disease or coeliac disease confirmed by biopsy
* Gastrointestinal malignancy
* Unable to comply with dietary restrictions required for the study.

Ages: 12 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 12 (Actual)
Dates: Start 2019-09-03 (Actual); Primary Completion 2020-10-29 (Actual); Study Completion 2020-10-29 (Actual)

PRIMARY OUTCOMES:
Oro-caecal Transit Time | 1 day of scanning
  Time taken after eating for ingested food to be identifiable at the caecum on MRI

SECONDARY OUTCOMES:
Gastric volume | 1 day of scanning
  Volume of stomach at each time point of digestion to measure gastric emptying time
Small bowel water content (corrected for body surface area) | 1 day of scanning
  Volume of water content in small bowel representing secretions and post prandial change in small bowel water content at T240 and T300
Colonic volume (corrected for body surface area) | 1 day of scanning
  Volume of colon representing ease of chyme passage through colon
Gastrointestinal symptoms | 1 day of scanning
  Gastrointestinal symptoms measured by patient reported outcomes to monitor relationships with outcomes measure by MRI

OTHER OUTCOMES:
Sigmoid colon volume | 1 day of scanning
  Volume of sigmoid colon
T1 relaxation of ascending colon chyme | 1 day of scanning
  An approximate measure of water content in chyme present in the ascending colon
Fat fraction of ascending colon chyme | 1 day of scanning
  A measure of fat content in chyme present in the ascending colon
Faecal elastase | 1 day
  A measure of elastase in stool to evaluate pancreatic function
Sputum and faecal microbiome | 1 day
  A measure of microbiome in sputum and stool
Faecal calprotectin | 1 day
  A measure of intestinal inflammation
Terminal Ileum motility | 1 day
  A measure of motility at the terminal ileum using the GIQuant tool in arbitrary units

CONTACTS AND LOCATIONS:
Overall Officials: Alan Smyth, Prof, Principal Investigator — University of Nottingham; Giles Major, Dr, Principal Investigator — University of Nottingham
Locations (1):
- Nottingham University Hospitals NHS Trust, Nottingham, Nottinghamshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
The data can be obtained by reasonable request to the study Principal Investigator and corresponding author Professor Alan Smyth (alan.smyth@nottingham.ac.uk) This will be assessed on a case-by-case basis. Applications should state the research question being addressed and include a link to the researcher's published protocol. This will be reviewed by the research team and a final decision to share data the responsibility of the Principal Investigator.

REFERENCES:
- [Derived] Ng C, Dellschaft NS, Hoad C, Marciani L, Spiller R, Crooks C, Hill T, Menys A, Mainz JG, Barr H, Gowland PA, Major G, Smyth AR. A randomised crossover trial of tezacaftor-ivacaftor for gut dysfunction in cystic fibrosis with magnetic resonance imaging (MRI) outcomes: a pilot study. NIHR Open Res. 2024 Mar 19;3:65. doi: 10.3310/nihropenres.13510.2. eCollection 2023. PMID 39139270